CLINICAL TRIAL: NCT00404495
Title: Phase 2 Single-Arm, Open Label Study Of Irinotecan In Combination With Temozolomide In Children With Recurrent Or Refractory Medulloblastoma And In Children With Newly Diagnosed High-Grade Glioma.
Brief Title: Combination of Irinotecan and Temozolomide in Children With Brain Tumors.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5961166
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Glioma; Medulloblastoma
MeSH Terms: conditions — Glioma; Medulloblastoma | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide + Irinotecan (Experimental)
  Interventions: Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 10 mg/m^2 per day on days 1-5 and days 8-12 in repeated 3 week cycles
Drug: Temozolomide — Temozolomide 100-125 mg/m^2 daily on days 1-5 in repeated 3 week cycles

SUMMARY:
This study will assess the rate of objective confirmed tumor response of irinotecan in combination with temozolomide in children with recurrent or refractory medulloblastoma and in children with newly diagnosed high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Recurrent or refractory medulloblastoma in which current standard treatment approaches have failed; biopsy is not required for recurrent disease.
* Cohort 2: Newly-diagnosed high-grade glioma (World Health Organization [WHO] grade 3 or 4)
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Diagnosis of brainstem glioma
* Concurrent administration of any other anti-tumor therapy
* Pre-existing uncontrolled diarrhea

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Australia (3):
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Parkville, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Denmark (2):
  - Pfizer Investigational Site, Aarhus N
  - Pfizer Investigational Site, Koebenhavn OE
- France (7):
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Villejuif
- Pfizer Investigational Site, Padua, Italy
- Pfizer Investigational Site, Warsaw, Poland
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Esplugues de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, El Palmar, Murcia
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- United Kingdom (7):
  - Pfizer Investigational Site, Soouthampton, Hampshire
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Sutton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5961166&StudyName=Combination%20of%20Irinotecan%20and%20Temozolomide%20in%20Children%20with%20Brain%20Tumors.

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide + Irinotecan for Medulloblastoma: For participants with medulloblastoma: Irinotecan 10 mg/m^2/day on Days 1-5 and Days 8-12 in repeated 3-week cycles. Temozolomide 100-125 mg/m^2 daily on Days 1-5 in repeated 3-week cycles; treatment duration: up to 1 year or until progression.
- Temozolomide + Irinotecan for High-Grade Glioma: For participants with high-grade glioma: Irinotecan 10 mg/m^2/day on Days 1-5 and Days 8-12 in repeated 3-week cycles. Temozolomide 100-125 mg/m^2 daily on Days 1-5 in repeated 3-week cycles; treatment duration: 2 cycles as a window phase before starting standard therapy.
Period: Overall Study
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Started | 66 | 17
Completed | 22 | 6
Not Completed | 44 | 11
Not completed — Death | 37 | 11
Not completed — Lost to Follow-up | 5 | 0
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma | Total
Number analyzed (Participants) | 66 | 17 | 83
Age, Customized [Number; unit: participants]
  2 years to 12 years | 49 | 12 | 61
  >12 years to 18 years | 17 | 5 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 3 | 24
  Male | 45 | 14 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response of Complete Response or Partial Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR). CR persisted on repeat imaging study at least (≥) 4 weeks after initial documentation of response. PR, for bidimensionally measurable disease, was a decrease by ≥50% of the sum of the products of the largest perpendicular diameters of all measurable lesions as determined by 2 observations not less than 4 weeks apart. Best overall response recorded any time while the participant was receiving treatment. External Response Review Committee (ERRC) assessment.
Time Frame: Baseline to 1 Year (medulloblastoma), Baseline to 6 Weeks (high-grade glioma)
Population: Primary Evaluable Population: subset of evaluable population predetermined by 2-stage Optimum Simon design. Medulloblastoma cohort: n=consecutive evaluable participants up to 46 if 6 responses obtained in first 15 evaluable participants. Glioma cohort: n=consecutive evaluable participants up to 29 if 1 response in first 10 evaluable participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 46 | 10
percentage of participants | 32.6 [19.5 to 48.0] | 0 [0 to 30.8]

2. Secondary Outcome: Percentage of Participants With Objective Response of Complete Response or Partial Response, Investigator's Assessment
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR. CR persisted on repeat imaging study ≥4 weeks after initial documentation of response. PR, in case of bidimensionally measurable disease, was a decrease by ≥50% of the sum of the products of the largest perpendicular diameters of all measurable lesions as determined by 2 observations not less than 4 weeks apart. Best overall response could be recorded any time while the participant was receiving treatment. Investigator's assessment.
Time Frame: Baseline to 1 Year (medulloblastoma), Baseline to 6 Weeks (high-grade glioma)
Population: Evaluable local population: Participants received at least 1 dose of study medication, had measurable disease under study, at least 1 on-study objective tumor assessment, completed at least 2 cycles of study treatment or progressed. Based on investigator's assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 63 | 17
percentage of participants | 34.9 [23.3 to 48.0] | 11.8 [1.5 to 36.4]

3. Secondary Outcome: Duration of Response
Description: Median duration (50%) of tumor response for participants with objective disease response: who have not progressed or died due to any cause; with a response and subsequent progression or death due to any cause for duration of response (DR). DR was defined as time from start of first documented objective tumor response (CR or PR) to first documented objective tumor progression or death due to any cause, whichever occurred first. DR (calculated in Weeks) = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7. Investigator's assessment.
Time Frame: Baseline to Date of Tumor Response (Up to 1 Year)
Population: Evaluable local population. Number of participants analyzed=number of participants who responded.
Measure: Median (Full Range); unit: weeks
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 22 | 2
weeks | 22.4 [6.9 to 46.6] | 36.3 [4.0 to 68.6]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from the date of first dose of study treatment to the date of the first documentation of progressive disease (PD), the date of treatment discontinuation except completion of treatment, or date of death due to cancer. Investigator's assessment.
Time Frame: Baseline to Date of Treatment Failure (Up to 1 Year)
Population: Evaluable local population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 63 | 17
months | 3.8 [2.9 to 5.4] | 1.6 [1.3 to 2.4]

5. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time in months from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever came first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7 multiplied by 4.33. Tumor progression was determined from oncologic assessment data (where data met the criteria for PD). Investigator's assessment.
Time Frame: Baseline to Date of Progression (Up to 1 Year)
Population: Evaluable local population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 63 | 17
months | 5.6 [3.8 to 7.4] | 1.6 [1.3 to 7.5]

6. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7 multiplied by 4.33. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death). Investigator's assessment.
Time Frame: Baseline to Date of Death (Up to 1 Year After Treatment)
Population: All participants. One participant in the Temozolomide + Irinotecan for Medulloblastoma cohort did not have recurrent or refractory medulloblastoma and 3 participants in the Temozolomide + Irinotecan for High-Grade Glioma cohort did not have high-grade glioma, and were not considered evaluable for survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Number analyzed (Participants) | 65 | 14
months | 16.7 [13.3 to 19.8] | 9.4 [5.8 to 20.2]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Temozolomide + Irinotecan for Medulloblastoma | Temozolomide + Irinotecan for High-Grade Glioma
Serious Adverse Events (participants affected / at risk) | 31/66 | 5/17
Other Adverse Events (participants affected / at risk) | 64/66 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide + Irinotecan for Medulloblastoma (N=66) | Temozolomide + Irinotecan for High-Grade Glioma (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 0
Blood culture positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coma (Nervous system disorders) | 3 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hydrocephalus (Nervous system disorders) | 3 | 1
Hypotonia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide + Irinotecan for Medulloblastoma (N=66) | Temozolomide + Irinotecan for High-Grade Glioma (N=17)
Anaemia (Blood and lymphatic system disorders) | 10 | 1
Eosinopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 10 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear canal erythema (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 5 | 1
Diplopia (Eye disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 3 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 22 | 4
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1
Anal erosion (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 23 | 4
Diarrhoea (Gastrointestinal disorders) | 38 | 10
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 7
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 3 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 42 | 13
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 6 | 2
Catheter site pain (General disorders) | 2 | 0
Catheter site rash (General disorders) | 2 | 0
Catheter site swelling (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Device occlusion (General disorders) | 1 | 0
Fatigue (General disorders) | 15 | 4
Feeling abnormal (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 14 | 2
Xerosis (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 3
Oral candidiasis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 0
Urinary tract infection (Infections and infestations) | 5 | 2
Viral infection (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 1
Aspartate aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood bicarbonate increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood culture positive (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood urea decreased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Heart rate (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Protein total increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 6 | 0
Weight increased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 5 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 4 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 20 | 5
Hydrocephalus (Nervous system disorders) | 3 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 4 | 0
Meningeal disorder (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Reflexes abnormal (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 5 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Tardive dyskinesia (Nervous system disorders) | 1 | 0
Tonic convulsion (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 4 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study had one treatment arm but two distinct cohorts with different diagnostics and treatment durations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.